CLINICAL TRIAL: NCT03688139
Title: Positive Valence System Function and Reward Exposure Therapy for Late-Life Depression
Brief Title: Reward Function and Therapy for Late-Life Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1803019076; K23MH116105 (NIH)
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Results first posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder
Keywords: depression; major depressive disorder; mental health; mood disorder; geriatric; late-life
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Psychological Well-Being; Mood Disorders | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Engage Therapy (Experimental): Participants receive Engage therapy for 9 weeks.
  Interventions: Behavioral: Engage Therapy
- Supportive Therapy (Active Comparator): Participants receive supportive therapy for 9 weeks.
  Interventions: Behavioral: Supportive Therapy

INTERVENTIONS:
Behavioral: Engage Therapy — Engage therapy is designed to help individuals with depression become involved in activities they previously enjoyed but have not been participating in since developing depression. In Engage therapy, individuals with depression work with a therapist to develop "action plans" to pursue rewarding activities of their choice.
  Arms: Engage Therapy
Behavioral: Supportive Therapy — Supportive therapy is designed to provide a warm and supportive environment in which individuals with depression can feel comfortable expressing their thoughts and feelings. In supportive therapy, therapists help patients identify themes in their thinking, provide reassurance, emphasize coping skills, and provide guidance as needed.
  Arms: Supportive Therapy

SUMMARY:
The goal of this study is to learn about changes in the brain that occur during Engage, a psychotherapy for depression in older adults, and how they may differ from changes that occur during supportive therapy. Older adults with depression will receive 9 weeks of either Engage or supportive therapy and will complete research assessments before the therapy begins and at weeks 3, 6, and 9 of treatment. Research assessments will include questionnaires, computer tasks, and recordings of electrical brain activity (also called electroencephalography or EEG).

DETAILED DESCRIPTION:
Late-life depression is prevalent and devastating, and response rates to even the most effective treatments are low. Outcomes may be improved by developing targeted interventions such as Engage - a new, easily disseminated, neurobiologically informed psychotherapy for late-life depression designed to restore impaired function of neural reward systems. This study will use event-related potentials and a panel of other reward system measures to assess target engagement in depressed older adults receiving Engage therapy, with a comparison group of depressed peers receiving supportive therapy. Participants will be randomly assigned to either Engage or supportive therapy and will complete research assessments at baseline and weeks 3, 6, and 9 (end of treatment).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 60 years.
* Diagnosis of unipolar major depressive disorder without psychotic features, determined by Structured Clinical Interview for the Diagnostic and Statistical Manual for Mental Disorders (SCID).
* Montgomery-Asberg Depression Rating Scale (MADRS) score greater than or equal to 20.
* Mini Mental State Exam (MMSE) score greater than or equal to 24.
* Off antidepressants or on a stable dose of an antidepressant for 12 weeks and no intent to change the dose in the next 10 weeks.
* Capacity to provide written consent for both research assessment and treatment.

Exclusion Criteria:

* Intent or plan to attempt suicide in the near future.
* Presence of current psychiatric diagnoses other than major depressive disorder without psychotic features, generalized anxiety disorder, or specific phobia.
* History of past psychiatric diagnoses other than major depressive disorder without psychotic features or anxiety disorders (separation anxiety disorder, specific phobia, social phobia, panic disorder, agoraphobia, or generalized anxiety disorder).
* Use of psychotropic drugs or cholinesterase inhibitors other than use of less than or equal to 0.5 mg of lorazepam daily up to five times per week.
* Neurological disorders (dementias, history of stroke, multiple sclerosis, Parkinson's disease, epilepsy, etc.); cardiac, renal, or respiratory failure; severe chronic obstructive pulmonary disease; metastatic cancer; or debilitated states or less common medical illnesses that may either influence neural systems of interest or ability to participate in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Bress, PhD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, White Plains, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The data collected during this study will be made available to other researchers after the main results have been published. To ensure data and participant security, we will make the data available to users under a data-sharing agreement.
Time Frame: The data will be made available after the main results have been published.
Access Criteria: Researchers interested in accessing the data will be asked to provide to the PI, and to the ALACRITY center with which the PI is affiliated, a proposal of hypotheses, variables needed to test these hypotheses, and plans for dissemination of findings. Before researchers are granted access, they will be asked to indicate in a signed document: 1) a commitment to using the data only for research purposes; 2) a plan for securing the data; 3) an agreement to either destroy or return the data once analyses are completed; and 4) and agreement not to share data with other users and to direct all such requests to the PI.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through community referrals, physical ads posted in locations frequented by older adults, a depression screening hotline maintained by the Weill Cornell Institute of Geriatric Psychiatry, and via ads posted on social media. The first participant was enrolled on 3/14/2019, and the last participant was enrolled on 9/26/2023.
Period: Overall Study
Arm/Group | Engage Therapy | Supportive Therapy
Started | 32 | 33
Completed | 28 | 29
Not Completed | 4 | 4
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Engage Therapy | Supportive Therapy | Total
Number analyzed (Participants) | 32 | 33 | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.79 (6.34) | 72.75 (7.64) | 70.31 (7.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 49
  Male | 7 | 9 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 31 | 33 | 64
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 27 | 29 | 56
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 33 | 65
Late Positive Potential [Mean (Standard Deviation); unit: microvolts] — The late positive potential (LPP) is an electroencephalographic (EEG)-derived measure of emotional engagement with positively valanced images. Population: Two participants dropped out before baseline and some data points are missing due to poor data quality or missed study assessments.
  microvolts
    number analyzed (Participants) | 29 | 32 | 61
    (all) | 4.84 (3.13) | 6.78 (4.87) | 5.86 (4.22)
Reward Positivity [Mean (Standard Deviation); unit: microvolts] — The reward positivity (RewP) is an electroencephalographic (EEG)-derived response to rewarding feedback from a guessing task. Population: Two participants dropped out before baseline and some data points are missing due to poor data quality or missed study assessments.
  microvolts
    number analyzed (Participants) | 28 | 29 | 57
    (all) | 2.15 (2.37) | 2.26 (3.80) | 2.21 (3.15)
P1 [Mean (Standard Deviation); unit: microvolts] — The P1 is an electroencephalographic (EEG)-derived measure of early visual attention that is elicited by visual stimuli. Population: Two participants dropped out before baseline and some data points are missing due to poor data quality or missed study assessments.
  microvolts
    number analyzed (Participants) | 29 | 32 | 61
    (all) | 1.92 (3.80) | 2.41 (3.09) | 2.18 (3.42)
Behavioral Activation [Mean (Standard Deviation); unit: units on a scale] — Behavioral activation will be measured using the Behavioral Activation for Depression Scale (BADS), a 25-item measure of behaviors targeted in behavioral activation therapies such as Engage. Scores range from 0 to 150, where higher scores on this measure indicate more participation in activities and social interactions, and lower scores indicate more social isolation, rumination, and avoidance of activities. Population: Two participants dropped out before baseline and some data points are missing due to missed study assessments.
  units on a scale
    number analyzed (Participants) | 29 | 32 | 61
    (all) | 82.72 (21.52) | 77.75 (15.77) | 80.11 (18.73)
Anhedonia [Mean (Standard Deviation); unit: units on a scale] — Anhedonia will be measured by the clinician-rated Snaith-Hamilton Pleasure Scale (SHAPS-C). The SHAPS-C measures pleasure and enjoyment experienced in response to a variety of situations. Scores range from 14 to 56, where higher scores indicate greater severity of anhedonia and lower scores indicate lower severity of anhedonia. Population: Two participants dropped out before baseline and some data points are missing due to missed study assessments.
  units on a scale
    number analyzed (Participants) | 30 | 32 | 62
    (all) | 30.30 (6.91) | 32.31 (6.35) | 31.34 (6.65)

OUTCOME MEASURES:

1. Primary Outcome: Change in Late Positive Potential to Rewarding Stimuli
Description: The late positive potential (LPP) is an electroencephalographic (EEG)-derived measure of emotional engagement with positively valanced images.
Time Frame: Change from baseline to week 9
Population: Two participants dropped out before baseline and some data points are missing due to poor data quality or missed study assessments.
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Engage Therapy | Supportive Therapy
Number analyzed (Participants) | 25 | 23
microvolts | 0.80 (3.24) | 0.07 (3.25)
Statistical Analysis 1: Comparison: Engage Therapy vs Supportive Therapy; Test type: Superiority; p = .08, Mixed Models Analysis; difference in slopes = 0.23
Statistical Analysis 2: Comparison: Engage Therapy; Test type: Other — This analysis tested whether the course of LPP was associated with the course of BADS over the 9-week treatment period in the Engage group; p = .14, Mixed Models Analysis; Slope = .03

2. Primary Outcome: Change in the Reward Positivity
Description: The reward positivity (RewP) is an electroencephalographic (EEG)-derived response to rewarding feedback from a guessing task.
Time Frame: Change from baseline to week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Engage Therapy | Supportive Therapy
Number analyzed (Participants) | 24 | 22
microvolts | -0.46 (3.66) | -0.60 (4.85)
Statistical Analysis 1: Comparison: Engage Therapy vs Supportive Therapy; Test type: Superiority; p = .69, Mixed Models Analysis; difference in slopes = -.06

3. Primary Outcome: Change in P1
Description: The P1 is an electroencephalographic (EEG)-derived measure of early visual attention that is elicited by visual stimuli.
Time Frame: Change from baseline to week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microvolts
Arm/Group | Engage Therapy | Supportive Therapy
Number analyzed (Participants) | 25 | 23
microvolts | -0.24 (1.39) | 0.43 (1.61)
Statistical Analysis 1: Comparison: Engage Therapy vs Supportive Therapy; Test type: Superiority; p = .69, Mixed Models Analysis; difference in slopes = -.03

4. Primary Outcome: Change in Behavioral Activation
Description: Behavioral activation will be measured using the Behavioral Activation for Depression Scale (BADS), a 25-item measure of behaviors targeted in behavioral activation therapies such as Engage. Scores range from 0 to 150, where higher scores on this measure indicate more participation in activities and social interactions, and lower scores indicate more social isolation, rumination, and avoidance of activities.
Time Frame: Change from baseline to week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage Therapy | Supportive Therapy
Number analyzed (Participants) | 26 | 28
units on a scale | 12.88 (14.64) | 18.93 (23.51)
Statistical Analysis 1: Comparison: Engage Therapy vs Supportive Therapy; Test type: Superiority; p = .39, Mixed Models Analysis; difference in slopes = -0.45

5. Secondary Outcome: Change in Anhedonia
Description: Anhedonia will be measured by the clinician-rated Snaith-Hamilton Pleasure Scale (SHAPS-C). The SHAPS-C measures pleasure and enjoyment experienced in response to a variety of situations. Scores range from 14 to 56, where higher scores indicate greater severity of anhedonia and lower scores indicate lower severity of anhedonia.
Time Frame: Change from baseline to week 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engage Therapy | Supportive Therapy
Number analyzed (Participants) | 27 | 28
units on a scale | -3.37 (5.96) | -2.07 (6.13)
Statistical Analysis 1: Comparison: Engage Therapy vs Supportive Therapy; Test type: Other — This analysis tested the hypothesis that change in LPP for each assessment interval would predict severity of anhedonia at the next assessment in Engage but not in Supportive Therapy; p = .58, Mixed Models Analysis; difference in slopes = -.10
Statistical Analysis 2: Comparison: Engage Therapy vs Supportive Therapy; Test type: Other — This analysis tested the hypothesis that change in SHAPS for each assessment interval would predict severity of anhedonia at the next assessment in Engage but not in Supportive Therapy; p = .96, Mixed Models Analysis; difference in slopes = .00

ADVERSE EVENTS:
Time Frame: Baseline to week 9 of study participation
Arm/Group | Engage Therapy | Supportive Therapy
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/33
Other Adverse Events (participants affected / at risk) | 1/32 | 7/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Engage Therapy (N=32) | Supportive Therapy (N=33)
Fall resulting in injury (General disorders) | 0 | 3
Leg pain requiring surgery (Musculoskeletal and connective tissue disorders) | 0 | 1
Abdominal and thoracic pain requiring endoscopy (Gastrointestinal disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Fractured pelvis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hair loss at EEG electrode site (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03688139/Prot_SAP_000.pdf